CLINICAL TRIAL: NCT00722748
Title: The Genebank at Scripps Clinic Registry
Brief Title: Genomic Investigation of Cardiovascular Diseases
Status: Active, not recruiting | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute, Scripps Translational Science Institute
Other Study IDs: HSC004714
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Atrial Fibrillation; Aortic Stenosis; Mitral Regurgitation; Idiopathic Cardiomyopathy
Keywords: Genebank; Gene registry; Cardiac Arrythmia Disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Atrial Fibrillation; Aortic Valve Stenosis; Mitral Valve Insufficiency; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cardiac Catheterization Patients
  Blood will be collected from the patients that will undergo heart catheterization for establishing a gene bank registry. Informed consent will take place prior to cardiac catheterization. 38 cc of blood collected will be processed to create a repository of DNA, RNA, and lymphoblastoid cell-line immortalization on selected patient populations, plasma and serum. The DNA will be amplified in certain patient populations to preserve the quantity.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Genebank: By creating a genebank from patient's blood donations we will ultimately be able to define genes for various cardiovascular conditions.

SUMMARY:
This proposal puts forward a research plan to initiate a genetic databank, henceforth referred to as The Genebank at Scripps Clinic Registry. This database will usher in genomic research at Scripps as we strive to stay at the forefront of cardiovascular research in the new century. Human subject donation allows for the creation of the proposed genebank.

DETAILED DESCRIPTION:
The completion of the human genome project within the final months of the previous millennium, is a landmark of scientific accomplishment. This achievement heralds the importance human and molecular genetics will play in the coming century in medicine. In short, one expects that dissecting the phenotypic aspects of disease to a culprit mutation/variation of a gene or collection of genes, will modify and or augment our present diagnostic ability leading on to new therapeutic interventions that are targeted based on these discoveries.

The broad application of human genetics will progress from the study of rare mendelian traits with complete penetrance compiled over the last 3-4 decades to a large number of "common" diseases that have multi-gene etiology with variable penetrance such as non-insulin dependent diabetes mellitus and hypertension. Cardiology will probably stay at a forefront of this transformation, as cardiovascular diseases (CVD) remain the major source of morbidity and mortality in developing countries, and is fast reaching the same status in the underdeveloped countries. Furthermore, the track record of rapid adaptation of new technology and research in the field of cardiology, would give further impetus to this transition. In the midst of these dynamic currents, this proposal puts forward a research plan to initiate a genetic databank, henceforth referred to as The Genebank at Scripps Clinic Registry. This database will usher in genomic research at Scripps as we strive to stay at the forefront of cardiovascular research in the new century.

The objective of this study is, to obtain blood samples in order to define genes for various cardiovascular conditions. The blood samples will go through DNA analysis and noted for 1 million SNP's per individual.

ELIGIBILITY:
Inclusion Criteria:

Candidates for this study must meet ALL of the following criteria:

* Age 18 years or older
* Be reliable, cooperative and willing to comply with all protocol-specified procedures and sub-study if consented.
* Able to understand and grant informed consent
* Have at least one of the following (a-g):

  1. Coronary Artery Disease (defined as):

     * Coronary artery bypass surgery or
     * Lesion >70% on cardiac or CT angiogram or
     * Percutaneous Coronary Intervention
  2. Myocardial infarction (defined as):

     * Diagnosed by elevated troponin level or
     * Diagnosed by ST segment elevations on EKG or
     * Diagnosed by pathologic Q waves on EKG or
     * Documented in the medical record or by self report
  3. Atrial Fibrillation (defined as):

     * Lone Atrial fibrillation (paroxysmal, persistent or permanent); OR
     * Lone Atrial Flutter (paroxysmal, persistent or permanent)
  4. Automatic Internal Cardiac Defibrillator
  5. Aortic Stenosis (defined by):

     * Calculated Aortic Valve Area ≤ 1.0 cm² or
     * Mean Pressure Gradient ≥ 40 mmHg or
     * Peak Pressure Gradient ≥ 64 mmHg or
     * Dimensionless Index < .25 or
     * Prior or planned Aortic Valve Replacement for Aortic Stenosis
  6. Mitral Regurgitation (insufficiency) (defined as)

     * Moderate to Severe (equivalent to +3 to +4) mitral regurgitation (insufficiency) on transthoracic echocardiogram as determined by the reading physician and structurally abnormal valve (i.e. myxomatous) and/or thickened or redundant leaflets; OR
     * Prior or planned Mitral Valve repair or replacement for mitral regurgitation
  7. Idiopathic (non-ischemic) Cardiomyopathy (defined as):

     * Diagnosed < age 40; OR
     * Non-ischemic etiology confirmed by cardiac angiography or CT angiography (may have non-obstructive or stable coronary artery disease if diagnosis of non-ischemic etiology of CM is established by cardiologist).

Exclusion Criteria:

Patients will be excluded if ANY of the following conditions apply:

* Previously enrolled in The Genebank at Scripps Clinic Registry
* Any active bleeding (i.e. GI bleed).
* Has a significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study
* Treatment with any investigational agents or devices within 30 days preceding enrollment in the study.
* Been administered or taken any CNS sedatives or depressants in the past 12 hours.
* Been administered or taken any CNS sedatives or depressants in the past 12 hours.
* Subject's qualifying diagnosis is Atrial fibrillation and they are known to have any one of the following:

  1. Prior myocardial infarction, coronary artery bypass surgery, or percutaneous coronary intervention
  2. EF < 45% at time of diagnosis (excluding tachycardia induced cardiomyopathy diagnosed by a cardiologist)
  3. Elevated left atrial pressures (> 20 mmHg)
  4. Dilated left atrium (> 4.0 cm or >2.0 cm/m2 body surface)
  5. Mitral valve disease with significant valve pathology

     * Mitral regurgitation/insufficiency greater than trace to mild on echo as determined by reading physician
     * Rheumatic mitral valve disease
  6. Congestive heart failure prior to diagnosis
  7. Hypertrophic cardiomyopathy
  8. Diagnosis following coronary artery bypass or valve replacement surgery
  9. Post heart transplant
  10. Congenital heart disease
  11. Diagnosed in setting of hyperthyroid
  12. COPD
  13. Obstructive sleep apnea
* Subject's qualifying diagnosis is Aortic Stenosis and they are known to have any one of the following:

  1. Bicuspid valve or other congenital abnormality of the aorta or aortic valve
  2. Evidence of Rheumatic involvement of the Aortic Valve
* Subject's qualifying diagnosis is Mitral regurgitation (insufficiency) and they are known to have any one of the following:

  1. Ejection fraction <50%
  2. Evidence of significant ischemic disease with regions of akinetic myocardium
  3. Rheumatic changes on echocardiogram (as determined by the reading physi4ian)

  5. Significant Mitral stenosis (greater than "mild" on echocardiogram as determined by the reading physician) 6. Evidence of valve perforation 7. Evidence of congenital abnormality (i.e. cleft valve)
* Subject's qualifying diagnosis is Idiopathic (non-ischemic) cardiomyopathy and they are known to have any one of the following:

  1. Ischemic cardiomyopathy
  2. Hypertrophic cardiomyopathy
  3. Viral cardiomyopathy
  4. Alcohol/drug induced cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from Scripps Health general diagnostic population, cardiology population, and outside referrals. Upon meeting the inclusion/exclusion criteria, each eligible patient will be given a consent form and the study will be discussed with them in a face-to-face discussion with the principal investigator, one of the co-investigators or one of the research coordinators. The patient (or legal representative) must sign the informed consent form prior to any study related procedures being performed.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2007-06; Primary Completion 2025-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
38 cc of blood obtained for DNA analysis. Medical information -diagnosis, disease history, medical treatments, response to treatments, laboratory tests, subject's age, ethnic background, and if available, related family history. | At the time of informed consent

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Topol, MD, Principal Investigator — Scripps Translational Science Institute
Locations (1):
- Scripps Health, La Jolla, California, United States

REFERENCES:
- See also: The webpage for Scripps Translational Science Institute — http://www.stsiweb.org